CLINICAL TRIAL: NCT00889187
Title: Phase I/II Study of Neoadjuvant Accelerated Short Course Radiation Therapy With Photons and Capecitabine for Resectable Pancreatic Cancer
Brief Title: Neoadjuvant Accelerated Short Course Radiation Therapy With Photons and Capecitabine for Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Excess toxicity was identified intraoperatively
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Harvey Mamon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-375
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Results first posted 2017-07-14 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Pancreatic Cancer
Keywords: radiation therapy; capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1 Cohort 1: Photon Rad (30 Gy/12 days)+Capecitabine (Experimental): Neoadjuvant Short-Course Photon Radiation:
  At dose level 1, a total dose of 30 Gy in 10 fractions (3 Gy/day) was prescribed to the 95% isodose and administered 5 days per week over 12 days.
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
  Interventions: Radiation: Neoadjuvant Short-Course Photon Radiation; Drug: Capecitabine
- Phase I Cohort 2: Photon Rad (25 Gy/11 days)+Capecitabine (Experimental): Neoadjuvant Short-Course Photon Radiation:
  At dose level 2, a total dose of 25 Gy in 5 fractions was prescribed to the 95% isodose and administered at 5 Gy per fraction over 11 days.
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
  Interventions: Radiation: Neoadjuvant Short-Course Photon Radiation; Drug: Capecitabine
- Phase I Cohort 3: Photon Rad (25 Gy/5 days)+Capecitabine (Experimental): Neoadjuvant Short-Course Photon Radiation:
  At dose level 3, a total dose of 25 Gy in 5 fractions was prescribed to the 95% isodose and administered at 5 Gy per fraction over 5 days.
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
  Interventions: Radiation: Neoadjuvant Short-Course Photon Radiation; Drug: Capecitabine
- All Phase I: Photon Rad+Capecitabine (Experimental): Neoadjuvant Short-Course Photon Radiation:
  All Phase I participants received the radiation regimen according to the established dose escalation schedule.
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
  Interventions: Radiation: Neoadjuvant Short-Course Photon Radiation; Drug: Capecitabine
- Phase II: Photon Rad (MTD)+Capecitabine (Experimental): Neoadjuvant Short-Course Photon Radiation:
  Phase II participants received the radiation regimen established in the Phase I study (MTD).
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
  Interventions: Radiation: Neoadjuvant Short-Course Photon Radiation; Drug: Capecitabine

INTERVENTIONS:
Radiation: Neoadjuvant Short-Course Photon Radiation
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
The purpose of this research study is to determine if it is possible to deliver high dose radiation in one week while also giving the drug capecitabine for the treatment of pancreatic cancer prior to surgery, to determine if this treatment can be given safely for the treatment of pancreatic cancer prior to surgery and, to determine if this treatment can improve the local control pancreatic cancer prior to surgery compared to historical controls of standard treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Phase I: To determine the feasibility and tolerability of radiation therapy for pancreatic cancer delivered with high dose external beam radiation in a one week accelerated schedule with concurrent capecitabine
* Phase II: To demonstrate a grade 3 or greater (any) toxicity rate of less than 20%

Secondary

* To determine local control and recurrence patterns of pancreatic cancer relative to a standard regimen of 50.4 Gy as seen in historical controls
* To determine the pathologic response rate
* To determine the progression-free survival
* To determine the surgical morbidity
* To determine 30-day post-operative mortality after pancreatic resection

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histologic proof of pancreatic ductal carcinoma is required prior to treatment.
* No evidence of metastatic disease as determined by chest CT scan, abdominal CT scan (or MRI with gadolinium and/or manganese), and all patients must be staged with a physical exam, chest CT, and abdominal CT with intravenous contrast.
* Only potentially resectable patients are eligible. Potentially resectable is defined as: a)no extrapancreatic disease, b)no evidence (on CT) of involvement of the celiac axis or superior mesenteric artery, and c)no evidence (on CT or MRI) of occlusion of the superior mesenteric vein or superior mesenteric-portal venous confluence.
* 18 years of age or older
* ECOG Performance status of 0 or 1
* Women of child bearing potential must practice adequate contraception and to refrain from breast feeding. Female patients must have a negative pregnancy test within 7 days of treatment
* Lab values as specified in the protocol

Exclusion Criteria:

* Patients cannot have hepatic or peritoneal metastases detected by imaging or laparoscopy prior to chemoradiation
* Serious concomitant systemic disorders incompatible with the study, such as significant cardiac or pulmonary morbidity, or ongoing infection as manifested by fever
* Pregnant or lactating women
* Life expectancy < 3 months
* Serious, uncontrolled, concurrent infection(s)
* Any prior chemotherapy or radiation for treatment of the patient's pancreatic tumor
* Treatment for other cancers within the last five years, except cured non-melanoma skin cancer and treated in situ cervical cancer
* Clinically significant cardiac disease or myocardial infarction within the last 12 months
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* Lack of physical integrity of the upper gastrointestinal tract or malabsorption syndrome
* Known, existing uncontrolled coagulopathy
* Unwillingness to participate or inability to comply with the protocol for the duration of the study
* Any prior fluoropyrimidine therapy (unless given in an adjuvant setting and completed at least 6 months earlier)
* Prior unanticipated severe reaction to fluoropyrimidine therapy, or known hypersensitivity to 5-fluorouracil or known DPD deficiency
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance or oral drug intake
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery
* Patients should not be on cimetidine as it can decrease the clearance of 5-FU. Another H2-blocker or proton pump inhibitor may be substituted before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2011-12-30 (Actual); Study Completion 2011-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Mamon, MD, PhD, Principal Investigator — Dana-Farber/Brigham and Women's Cancer Center
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Wo JY, Mamon HJ, Ferrone CR, Ryan DP, Blaszkowsky LS, Kwak EL, Tseng YD, Napolitano BN, Ancukiewicz M, Swanson RS, Lillemoe KD, Fernandez-del Castillo C, Hong TS. Phase I study of neoadjuvant accelerated short course radiation therapy with photons and capecitabine for resectable pancreatic cancer. Radiother Oncol. 2014 Jan;110(1):160-4. doi: 10.1016/j.radonc.2013.10.027. Epub 2013 Nov 11. PMID 24231241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from Dec 2009 and Sep 2011.
Period: Overall Study
Arm/Group | Phase 1 Cohort 1: Photon Rad (30 Gy/12 Days)+Capecitabine | Phase I Cohort 2: Photon Rad (25 Gy/11 Days)+Capecitabine | Phase I Cohort 3: Photon Rad (25 Gy/5 Days)+Capecitabine | Phase II: Photon Rad (MTD)+Capecitabine
Started | 3 | 3 | 4 | 0
Completed | 3 | 3 | 4 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Phase I: Photon Rad+Capecitabine
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 62.6 [57 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Neoadjuvant Short-Course Photon Radiation Therapy Maximum Tolerated Dose (MTD) [Phase I]
Description: Neoadjuvant short-course photon radiation therapy MTD in combination with capecitabine 825 mg/m2 orally BID for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If none of 3 initial patients or only 1 of 6 patients have a DLT on dose level 3 then 6 additional patients are treated at this dose. If during this expansion, the rate of DLT exceeds 30% then the next lower dose level is declared the MTD. If no DLTs are observed, the MTD is not reached.
Time Frame: within 3 weeks of the start of chemoradiation therapy
Population: The analysis dataset is comprised of all treated patients.
Measure: Number; unit: Gy per fraction
Arm/Group | All Phase I: Photon Rad+Capecitabine
Number analyzed (Participants) | 10
Gy per fraction | NA — The study was closed early due to unexpected intraoperative complications. No patients developed a pre-specified DLT in the 10 treated patients. The MTD was not established.

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: DLT occurring within 3 weeks of the start of chemoradiation therapy was defined as: Grade 3 non-hematologic or hematologic toxicity requiring interruption of >7 days (d) of chemo or >3d chemoradiation; Grade 4 non-hematologic; Grade 4 neutropenia or thrombocytopenia; Treatment-related death; Delays in surgery >3 weeks due to treatment-related toxicity. A 30% increase in any surgical complication rate beyond those previously established rates (readmission rate: 16%; pancreatic fistula/intra-abdominal abscess/infection rate: 27%, major intra-abdominal bleeding requiring return to OR: 1.6%, delayed gastric emptying: 4.4%, and superficial wound infection rate: 8%) was also considered a DLT.
Time Frame: within 3 weeks of the start of chemoradiation therapy
Population: The analysis dataset is comprised of all treated patients.
Measure: Number; unit: patients with DLT
Arm/Group | Phase 1 Cohort 1: Photon Rad (30 Gy/12 Days)+Capecitabine | Phase I Cohort 2: Photon Rad (25 Gy/11 Days)+Capecitabine | Phase I Cohort 3: Photon Rad (25 Gy/5 Days)+Capecitabine
Number analyzed (Participants) | 3 | 3 | 4
patients with DLT | 0 | 0 | 0

3. Primary Outcome: Grade 3-5 Toxicity Rate [Phase II]
Description: All Grade 3-5 events based on CTCAEv3 related to the accelerated dose (attribution possible, probable, definite) as reported on case report forms.
Time Frame: within 3 weeks of the start of chemoradiation therapy
Population: The study did not proceed to phase II due to unexpected intraoperative complications experienced by patients enrolled on phase I.
Groups:
- Experimental: Phase II: Photon Rad (MTD)+Capecitabine: Phase II participants received the radiation regimen established in the Phase I study (MTD).
  Chemotherapy:
  Capecitabine was given orally 825 mg/m2 BID (total 1650 mg/m2 per day) for ten consecutive weekdays, beginning on the morning of the first day of radiation therapy.
  Patients underwent resection of their pancreatic cancer 1-3 weeks after the completion of chemoradiation. It was recommended that patients undergoing R0 or R1 resections receive adjuvant treatment with 4-6 cycles of gemcitabine-based therapy per institutional policy, to start 4 to 10 weeks after the operation.
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

4. Secondary Outcome: Local Recurrence Rate [Phase II]
Description: Local recurrence rate is defined as the proportion of patients with evidence of tumor recurrence within the radiation field based on RECIST criteria. Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease was assessed radiologically at baseline and after treatment every 6 months for first 2 years and annually in years 3-5.
Population: as for outcome 3
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: Pathologic Response Rate [Phase II]
Description: Pathologic response rate is the proportion of patients with the pathologic specimen absent any viable tumor cell. Pathological review of the pancreaticoduodenectomy specimen will be performed according to the AJCC Staging Classification, 6th edition. Initial gross evaluation and identification of resection margins will be performed jointly by the surgeon and the pathologist.
Time Frame: Assessed after resection; Patients underwent resection of their pancreatic cancer up to 3 weeks after completion of chemoradiation therapy
Population: as for outcome 3
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression-Free Survival (PFS) [Phase II]
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. Patients alive whose disease had not progressed are censored at date of last disease evaluation
Time Frame: as for outcome 4
Population: as for outcome 3
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

7. Secondary Outcome: Surgical Morbidity Rate [Phase II]
Description: The proportion of patients experienced any grade 3-4 adverse event based on CTCAEv3 related to the surgery (attribution possible, probable, definite) as reported on case report forms.
Time Frame: as for outcome 5
Population: as for outcome 3
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

8. Secondary Outcome: Surgical Mortality Rate [Phase II]
Description: The proportion of patients with a death related to the surgery (CTCAEv3 attribution possible, probable, definite).
Time Frame: Assessed up to 30 days after resection; Patients underwent resection of their pancreatic cancer up to 3 weeks after completion of chemoradiation therapy
Population: as for outcome 3
Arm/Group | Experimental: Phase II: Photon Rad (MTD)+Capecitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed continuously up to 3 weeks from the start of chemoradiation therapy.
Description: Serious AEs: AE that results in death; is life-threatening; requires or prolongs inpatient hospitalization; is disabling; is a congenital anomaly or birth defect; is medically significant or requires medical or surgical intervention to prevent one of the above outcomes. Other AEs: Remaining AEs (maximum grade by toxicity type) without regard to treatment attribution.The hemorrhage/bleeding-other case was gastrointestinal (GI) hemorrhage; no further data is available to specify infection-other.
Arm/Group | Phase 1 Cohort 1: Photon Rad (30 Gy/12 Days)+Capecitabine | Phase I Cohort 2: Photon Rad (25 Gy/11 Days)+Capecitabine | Phase I Cohort 3: Photon Rad (25 Gy/5 Days)+Capecitabine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: Photon Rad (30 Gy/12 Days)+Capecitabine (N=3) | Phase I Cohort 2: Photon Rad (25 Gy/11 Days)+Capecitabine (N=3) | Phase I Cohort 3: Photon Rad (25 Gy/5 Days)+Capecitabine (N=4)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Lymphopenia (Investigations) | 1 | 0 | 0
Infection-Other (Infections and infestations) | 0 | 1 | 0
Hemorrhage/Bleeding-Other (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: Photon Rad (30 Gy/12 Days)+Capecitabine (N=3) | Phase I Cohort 2: Photon Rad (25 Gy/11 Days)+Capecitabine (N=3) | Phase I Cohort 3: Photon Rad (25 Gy/5 Days)+Capecitabine (N=4)
Abdomen, pain (Gastrointestinal disorders) | 1 | 2 | 2
Alkaline phosphatase (Investigations) | 1 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
ALT, SGPT (Investigations) | 1 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 3
AST, SGOT (Investigations) | 1 | 0 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Bilirubin (Investigations) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 1 | 0
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Fatigue (General disorders) | 1 | 3 | 3
Fever w/o neutropenia (General disorders) | 2 | 0 | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Leukocytes (Investigations) | 0 | 1 | 1
Lymphopenia (Investigations) | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 1 | 3 | 3
Pain-other (General disorders) | 0 | 1 | 0
Perforation, cecum (Gastrointestinal disorders) | 0 | 1 | 0
Platelets (Investigations) | 0 | 0 | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stomach, pain (Gastrointestinal disorders) | 0 | 1 | 0
Urine color (Renal and urinary disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 2
Weight loss (Investigations) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The study did not proceed to phase II due to unexpected intraoperative complications experienced by patients enrolled on phase I.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No